CLINICAL TRIAL: NCT07021573
Title: Protoporphyrin Imaging in Multispectral Evaluation of Resections
Acronym: PRIMER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: PRIMER
Record Dates: First submitted 2025-05-13; First posted 2025-06-15 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-05

CONDITIONS: Glioma
Keywords: Suspected high-grade gliomas
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Intervention Model Description: There are 2 groups: group 1 (GBM-like) includes patients with high-grade gliomas and significant contrast enhancement on preoperative MRI. Group 2 (LGG-like) will include patients with suspected HGG and little to no contrast enhancement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GMB like or LGG like (Other): There are 2 groups: group 1 (GBM-like) includes patients with high-grade gliomas and significant contrast enhancement on preoperative MRI. Group 2 (LGG-like) will include patients with suspected HGG and little to no contrast enhancement.
  Interventions: Device: KINEVO 900 S with BLUE 400

INTERVENTIONS:
Device: KINEVO 900 S with BLUE 400 — The investigational device consists of a CE marked (MDR) surgical microscope KINEVO 900 S by Carl Zeiss Meditec AG, including the BLUE 400 fluorescence option. This microscope is equipped with an additional component (CALLAO), provided by the Carl Zeiss Meditec AG, that allows for extended, multispectral, image acquisition in the operating room. CALLAO consists of an optical setup with additional cameras, that can be mounted on the main system KINEVO 900 S, and a second light source for specific illumination during image acquisition with the CALLAO cameras.
  Other Names: CALLAO

SUMMARY:
Observational non-interventional investigation to evaluate the potential of multispectral imaging in improving tumor visualization.

DETAILED DESCRIPTION:
The clinical study is conducted in the post-market stage according to ISO 14155 Annex I.1 as it is performed with a CE marked microscope system. An additional component (CALLAO) will be added to the microscope. The intended use of the microscope as well as the surgical procedure remain unchanged by this addition. CALLAO allows for taking pictures of the situs in the OR which increases the surgery duration by <1min per picture. Therefore, this is a non-interventional study with a minimal burden to subjects.

The clinical investigation is not for a conformity assessment purpose. The burden to subjects is non-interventional.

ELIGIBILITY:
Inclusion criteria:

* Age Requirement: Patients must be 18 years of age or older.
* Diagnosis: Patients with a preoperative diagnosis of a suspected high-grade glioma based demographics and MRI imaging.
* MRI Findings: Patients must meet one of the following criteria:

  * Group 1: Suspected high-grade glioma with contrast enhancement on MRI (GBM-like).
  * Group 2: Suspected high-grade glioma without contrast enhancement on MRI (LGG-like).
* Surgical Resection: Patients scheduled to undergo surgical resection of the tumor as part of standard treatment.
* 5-ALA Administration: Patients who will receive 5-aminolevulinic acid (5-ALA) for fluorescence guidance during surgery.
* Post-op MRI: Patients who are able to undergo pre- and postoperative MRI (standard of care at the center).
* Informed Consent: Patients who are able to understand and provide written informed consent prior to enrollment in the study.
* Eligibility for Multispectral Imaging: Patients whose surgical procedures allow for the use of multispectral imaging technology for tumor visualization.
* Performance Status: Patients with a Karnofsky Performance Status (KPS) of 60 or greater, indicating that they are capable of at least limited self-care.
* No Prior Treatment: Patients who have not received prior treatment for the current brain tumor, including surgery, radiotherapy, or chemotherapy.

Exclusion criteria:

* Patients with a known allergy or contraindication to 5-aminolevulinic acid (5-ALA) or its components.
* Use of all other fluorescent markers.
* Patients with a history of porphyria or other disorders related to 5-ALA metabolism.
* Patients with recurrent gliomas or those who have received prior treatment for their current brain tumor, including surgery, radiotherapy, or chemotherapy.
* Pregnant or breastfeeding patients, due to potential risks associated with 5-ALA administration.
* Patients with severe comorbidities or other medical conditions that, in the investigator's opinion, would pose an unacceptable risk or compromise the safety of participation in the study.
* Patients with a Karnofsky Performance Status (KPS) below 60, indicating an inability to perform minimal self-care.
* Patients with a history of severe hepatic or renal impairment that may impact the metabolism of 5-ALA.
* Patients unable to undergo MRI imaging for any reason (e.g., presence of non-MRI-compatible implants).
* Patients unable to provide written informed consent due to cognitive, language, or other barriers.
* Patients with tumors located in regions where fluorescence imaging is not technically feasible or where the use of multispectral imaging could interfere with the standard surgical approach.
* Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Primary objective | 12 months
  Detection of Tumor cells and fluorescence in biopsied tissue

SECONDARY OUTCOMES:
Secondary objectives | 12 months
  Correlation with Histopathology, Diagnostic Performance Metrics, Molecular or Cellular Characterization, Clinical Correlation, Imaging Technology Performance, Impact on Clinical Decision-Making

CONTACTS AND LOCATIONS:
Locations (10):
- Universitätsklinik für Neurochirurgie der Medizinischen Universität Innsbruck, Innsbruck, Austria
- Germany (7):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Freiburg - Klinik für Neurochirurgie im Neurozentrum, Freiburg im Breisgau
  - Universitätsklinikum Göttingen - Neurochirurgische Klinik, Göttingen
  - Klinik und Poliklinik für Neurochirurgie, LMU Klinikum München, München
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Universitätsklinikum Münster - Klinik für Neurochirurgie, Münster
  - Universitätsklinikum Tübingen, Universitätsklinik für Neurochirurgie, Tübingen
- Switzerland (2):
  - Inselspital Bern, Universitätsklinik für Neurochirurgie, Bern
  - Hôpitaux universitaires de Genève - NeuroCentre, Geneva

IPD SHARING:
Plan to Share IPD: No